CLINICAL TRIAL: NCT04684446
Title: A Phase I/II Single-Blinded Randomized Safety and Immunogenicity Study in Adults of AZD1222 and rAd26-S Administered as Heterologous Prime Boost Regimen for the Prevention of COVID 19
Brief Title: Study in Adults of AZD1222 and rAd26-S Administered as Heterologous Prime-Boost Regimen for the Prevention of COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: AstraZeneca (Industry); Russian Direct Investment Fund (Industry); The Gamaleya National Center of Epidemiology & Microbiology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D8111C00003
Record Dates: First submitted 2020-12-23; First posted 2020-12-24 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: COVID-19 Prevention; AZD1222 vaccine; rAd26-S; Sputnik V
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19; Gam-COVID-Vac vaccine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): AZD1222 on Day 1 followed by rAd26-S on Day 29
  Interventions: Biological: AZD1222
- Arm 2 (Experimental): rAd26-S on Day 1 followed by AZD1222 on Day 29
  Interventions: Biological: rAd26-S

INTERVENTIONS:
Biological: AZD1222 — Participants will receive 1 intramuscular (IM) injection of 5 ×1010 viral particles (vp) (nominal) of AZD1222 on Day 1 followed by rAd26-S 1×1011 viral particles (vp) (nominal) on Day 29 of the study
  Arms: Arm 1
Biological: rAd26-S — Participants will receive 1 IM injection of rAd26-S on Day 1 followed by AZD1222 on Day 29
  Other Names: Sputnik V
  Arms: Arm 2

SUMMARY:
The objective is to evaluate the safety and immunogenicity of AZD1222 given in combination with (either before or after) rAd26-S, for the prevention of COVID 19 in adults ≥ 18 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age at the time of signing the informed consent
2. Overtly healthy as determined by medical evaluation, or

   - Medically stable such that, according to the judgment of the investigator, hospitalisation within the study period is not anticipated and the participant appears likely to be able to remain in follow-up through the end of protocol-specified follow-up.

   o A stable medical condition is defined as disease not requiring significant change in therapy or hospitalisation for worsening disease during the 3 months prior to enrolment
3. Able to understand and comply with study requirements/procedures based on the assessment of the investigator
4. Reproduction:

Female participants

1. Women of childbearing potential must:

   * Have a negative pregnancy test on the day of screening and on Day 1
   * Use one highly effective form of birth control for at least 28 days prior to Day 1 and agree to continue using one highly effective form of birth control through 60 days following administration of the second dose of study vaccine. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly.

   Periodic abstinence, the rhythm method, and withdrawal are NOT acceptable methods of contraception.
2. Women are considered of childbearing potential unless they meet either of the following criteria:

   * Surgically sterilised (including bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or
   * Postmenopausal

     6. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

   Exclusion Criteria:

   Medical Conditions
   1. Known past laboratory-confirmed SARS-CoV-2 infection.
   2. Positive SARS-CoV-2 RT PCR test at screening.
   3. Seropositivity to SARS-CoV-2 at screening.
   4. Significant infection or other illness, including fever > 37.8°C on the day prior to or on the day of randomization 5. Thrombocytopenia ≥ Grade 2 (i.e. < 100 000/mm^3) 6. Clinically significant neutropenia (as determined by the investigator). 7. Clinically significant anaemia (as determined by the investigator) 8. Any confirmed or suspected immunosuppressive or immunodeficient state; including human immunodeficiency virus (HIV) infection; asplenia; recurrent severe infections and use of chronic immunosuppressant medication (within the past 6 months(≥ 20 mg/day of prednisone or its equivalent, given daily or on alternate days for ≥ 15 days within 30 days prior to vaccination), except topical/inhaled steroids or short-term oral steroids ( course lasting ≤ 14 days).

   9. History of allergy to any component of the vaccine 10. Any history of anaphylaxis or angioedema. 11. Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and uterine cervical carcinoma in situ).

   12. History of serious psychiatric condition likely to affect participation in the study.

   13. Bleeding disorder (eg, factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.

   14 Suspected or known current alcohol or drug dependency. 15 History of Guillan-Barré syndrome or any other demyelinating condition. 16 Any other significant disease, disorder or finding which may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study or impair interpretation of the study data.

   17 Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness (mild/moderate well controlled comorbidities are allowed).

   18. Prior splenectomy 19. History of cerebral venous sinus thrombosis or experienced major venous and/or arterial thrombosis.

   20. Receipt of any vaccine (licensed or investigational) other than the study intervention within 30 days before and after each study vaccination.

   21. Prior or planned receipt of an investigational or licensed vaccine or product likely to impact on interpretation of the trial data (eg, adenovirus vectored vaccines, any coronavirus vaccines).

   22. Administration of immunoglobulins and/or any blood products within the 3 months preceding the planned administration of the vaccine candidate.

   23. Continuous use of anticoagulants, such as coumarins and related anticoagulants (ie, warfarin) or novel oral anticoagulants (ie, apixaban, rivaroxaban, dabigatran and edoxaban).

   24. Participation in COVID-19 prophylactic drug trials for the duration of the study.

   25. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).

   26. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

   27. Previous randomisation in the present study 28. For female subjects only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.

   29. Unwilling to refrain from blood donation during the course of the study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Antibody seroconversion rate (≥ 4-fold increase from baseline) against SARS-CoV-2 neutralising antibodies 29 days post second vaccination. | Day 29 through Day 57
  Immunogenicity
Incidence of local and systemic solicited AEs for 7 days following each vaccination (Day 1 through Day 7 for first vaccination and Day 29 through Day 35 for second vaccination). | Day 1 through Day 7 and Day 29 through Day 35
  Safety
Incidence of unsolicited AEs, SAEs and AESIs through 29 days post each vaccination (ie, until Day 29 following the first vaccination and Day 57 following the second vaccination). | 57 days
  Safety

SECONDARY OUTCOMES:
Incidence of SAEs and AESIs after first vaccination until study end (Day 180). | 180 days
  Safety
Antibody seroconversion rate (≥ 4-fold increase from baseline) against SARS-CoV-2 Spike protein | 180 days
  Immunogenicity
Antibody seroconversion rate (≥ 4-fold increase from baseline) against RBD antigen. | 180 days
  Immunogenicity
GMT and GMFR of immunogenicity against Spike and RBD antigens (MSD serology assay) at the day of vaccination (baseline), Day 15, 29 days post each vaccination and at study end (Day 180). | 180 days
  Immunogenicity
Antibody seroconversion rate (≥ 4-fold increase from baseline) SARS-CoV-2 neutralising antibodies 29 days post first vaccination | Day 1 through Day 29
  Immunogenicity
GMT and GMFR of immunogenicity as measured by SARS-CoV-2 neutralising antibodies at day of vaccination (baseline), Day 15, 29 days post each vaccination and at study end (Day 180). | 180 days
  Immunogenicity
Intracellular cytokine staining, including quantification of Th1/Th2 responses, and flow cytometry for B- and T-cell responses from day of dosing baseline to 29 days post each vaccination and until study end | 180 days
  Safety
A binary response, whereby a participant is defined as a COVID-19 case if their illness (virologically confirmed [RT-PCR positive] and symptomatic) occurs | Day 29 through Day 180
  Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (4):
- Russia (4):
  - OJSC Clinical and Diagnostic Center Euromedservice, Moscow
  - LLC PiterClinica, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education " First Saint Petersburg State Medical University named after Academician I. P. Pavlov" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - Federal State Budget Institution "Scientific and Research Institute of Flu n.a. A.A. Smorodintseva" of Ministry of Health of Russian Federation, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home